CLINICAL TRIAL: NCT04630327
Title: Validation of the Russian and Kazakh Versions of the Beck Depression Inventory and Beck Anxiety Inventory Among Female Cancer Patients
Brief Title: Validation of the Russian and Kazakh Versions of the Beck Depression Inventory and Beck Anxiety Inventory
Status: Completed | Type: Observational
Sponsor: Kazakh Medical University of Continuing Education (Other)
Responsible Party: Sponsor
Other Study IDs: 06-2020/1
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Depression; Anxiety; Breast Cancer; Ovarian Cancer; Cervical Cancer; Lung Cancer; Colon Cancer
Keywords: depression; anxiety; breast cancer; validation study; female cancer patients
MeSH Terms: conditions — Depression; Anxiety Disorders; Breast Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Lung Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female Cancer Patients: Female cancer patients with no history of previously diagnosed depression or anxiety and who have been referred to or have been receiving treatment at Almaty Oncology Center or Kazakh Scientific Research Institute of Oncology and Radiology
  Interventions: Other: Beck Depression Inventory-21 (diagnostic survey); Other: Beck Anxiety Inventory; Other: Interview using The International Classification of Diseases in tenth edition (ICD-10) criteria

INTERVENTIONS:
Other: Beck Depression Inventory-21 (diagnostic survey) — Kazakh or Russian versions of the Beck Depression Inventory-21will be filled by female cancer patients
  Other Names: BDI-II
Other: Beck Anxiety Inventory — Kazakh or Russian versions of the Beck Anxiety Inventory will be filled by female cancer patients
  Other Names: BAI
Other: Interview using The International Classification of Diseases in tenth edition (ICD-10) criteria — Interview using The International Classification of Diseases in tenth edition (ICD-10) criteria as a gold standard of diagnosing depression or anxiety

SUMMARY:
Depression and anxiety in female patients with cancer are serious comorbidities that affect the quality of life for patients and their survival rates as they have poorer health outcomes. This validation study is a part of the study on the prevalence of depression and anxiety among breast cancer patients. This study aims to investigate the validity of the Kazakh and Russian versions of the Beck Depression Inventory (BDI-II) and Beck Anxiety Inventory (BAI) among female cancer patients in Almaty, Kazakhstan.

ELIGIBILITY:
Inclusion Criteria:

* adult female patients between 18 and 65 years of age with a primary diagnosis of breast cancer; ovarian cancer; cervical cancer; colon cancer; lung cancer;
* Russian or Kazakh language fluency;
* consent to participate;

Exclusion Criteria:

* history of diagnosed depression or anxiety;
* current use of antidepressants;
* referral to palliative care

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female cancer patients patients
Study Population: Adult female patients between 18 and 65 years of age with a primary diagnosis of breast cancer; ovarian cancer; cervical cancer; colon cancer; lung cancer; who have been referred to or have been receiving treatment at Almaty Oncology Center or Kazakh Scientific Research Institute of Oncology and Radiology
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
BDI-II Score at Baseline: | Baseline
  Beck Depression Inventory (BDI-II) Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represents a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.
BDI-II Score on day 14 | Day 14
  Beck Depression Inventory (BDI-II) Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represents a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.
BAI Score at Baseline | Baseline
  Beck Anxiety Inventory (BAI) is a 21-item self-reported questionnaire which measures the existenceand severity of symptoms of anxiety. Each of the 21 items on BAI tool represents an anxiety symptom. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and 26 - 63 as "Severe".
BAI Score Day 14 | Day 14
  Beck Anxiety Inventory (BAI) is a 21-item self-reported questionnaire which measures the existenceand severity of symptoms of anxiety. Each of the 21 items on BAI tool represents an anxiety symptom. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and 26 - 63 as "Severe".
ICD-10 diagnosis at baseline | Baseline
  The ICD-10 sets criteria for diagnosis of major depressive disorder and generalized anxiety disorder, and will be used as a gold standard of diagnosis of depression and anxiety.
ICD-10 diagnosis on Day 14 | Day 14
  The ICD-10 sets criteria for diagnosis of major depressive disorder and generalized anxiety disorder, and will be used as a gold standard of diagnosis of depression and anxiety.
Internal consistency of the BAI | Day 14
  Internal consistency of the subscales will be evaluated with Cronbach's alpha. Values between 0.70 and 0.90 will be considered good and greater than 0.90 will be considered excellent.
Internal consistency of the BDI-II | Day 14
  Internal consistency of the subscales will be evaluated with Cronbach's alpha. Values between 0.70 and 0.90 will be considered good and greater than 0.90 will be considered excellent.
Test - retest reliability of the BDI-II questtionaire | Day 14
  Test - retest reliability of the BDI-II questtionaire on Day 14. Test-retest reliability coefficients vary between 0 and 1, where:
  1 : perfect reliability,
  * 0.9: excellent reliability,
  * 0.8 < 0.9: good reliability,
  * 0.7 < 0.8: acceptable reliability,
  * 0.6 < 0.7: questionable reliability,
  * 0.5 < 0.6: poor reliability, < 0.5: unacceptable reliability, 0: no reliability. On this scale, a correlation of .9(90%) would indicate a very high correlation (good reliability) and a value of 10% a very low one (poor reliability).
Test - retest reliability of the BAI questtionaire | Day 14
  Test - retest reliability of the BAI questtionaire on Day 14. Test-retest reliability coefficients vary between 0 and 1, where:
  1 : perfect reliability,
  * 0.9: excellent reliability,
  * 0.8 < 0.9: good reliability,
  * 0.7 < 0.8: acceptable reliability,
  * 0.6 < 0.7: questionable reliability,
  * 0.5 < 0.6: poor reliability, < 0.5: unacceptable reliability, 0: no reliability. On this scale, a correlation of .9(90%) would indicate a very high correlation (good reliability) and a value of 10% a very low one (poor reliability).
Sensitivity and Specificity of the BDI-II at baseline | Baseline
  Sensitivity and Specificity of the BDI-II at baseline compared to ICD-10 criteria. Beck Depression Inventory (BDI-II) Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represents a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.
Sensitivity and Specificity of the BAI at baseline | Baseline
  Sensitivity and Specificity of the BAI at baseline compared to ICD-10 criteria. Beck Anxiety Inventory (BAI) is a 21-item self-reported questionnaire which measures the existenceand severity of symptoms of anxiety. Each of the 21 items on BAI tool represents an anxiety symptom. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and 26 - 63 as "Severe".

CONTACTS AND LOCATIONS:
Overall Officials: Botagoz Turdaliyeva, Professor, Study Director — Kazakh Medical University of Continuing Education
Locations (2):
- Kazakhstan (2):
  - Kazakh Scientific Research Institute of Oncology and Radiology, Almaty
  - Almaty Oncology Center, Almaty

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable IPD will be shared upon request with all required information
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available upon completion of the study primary analysis
Access Criteria: Only people with access will be able to see the data